CLINICAL TRIAL: NCT02662075
Title: Acute Effects of Electronic Cigarettes on Platelet, Vascular Endothelial Function, and Inflammation in Healthy Active Smokers
Brief Title: Effect of Electronic Cigarettes on Platelets, Endothelium and Inflammation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-02083
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Smoking
Keywords: alternative tobacco products (ATPs); electronic cigarettes
MeSH Terms: conditions — Smoking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E-cigarette/tobacco Smoking Exposure (Experimental)
  Interventions: Device: E-cigarette/tobacco Smoking Exposure

INTERVENTIONS:
Device: E-cigarette/tobacco Smoking Exposure — Subjects will be asked to smoke an e-cigarette containing the equivalence of nicotine in one tobacco cigarette (15 puffs) in the presence of research staff. Each puff will be timed at 4 seconds and there should be a 20-30 seconds interpuff interval as previously recommended.

SUMMARY:
The primary purpose of this study is to evaluate the acute effects of electronic cigarette (e-cigarette) smoking on measurable biomarkers of platelet function, vascular endothelial function and inflammation in healthy active smokers. 10 healthy subjects, smokers, with no other medical conditions will be included in this study and measurements will be obtained at baseline and after smoking an e-cigarette. The study will contribute to the understanding of the effects of e-cigarettes on cardiovascular physiology, specifically establishing if the use of e-cigarettes increases platelet aggregation and platelet activation when compared to baseline in healthy active smokers, if the use of e-cigarettes decreases brachial artery flow-mediated dilation compared to baseline in healthy active smokers, and to determine the association between biomarkers of inflammation, platelet function, and vascular endothelial function before and after use of e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Adult English speaking subjects able and willing to provide written informed consent
* Active tobacco cigarette smoker
* History of active smoking tobacco cigarettes for 3-10 years (at least 10 cigarettes per day). The rational for inclusion of active smokers is based on prior data showing that most e-cigarette users have smoked moderate to high amount of tobacco cigarettes in the past
* No other use of alternative tobacco or nicotine products
* No history of hypertension, diabetes, cardiovascular disease, stroke, peripheral arterial disease, asthma or other chronic lung disease.

Exclusion Criteria:

* Use of aspirin, clopidogrel, prasugrel, ticagrelor, warfarin, statins, colchicine, nitrates, steroids, fish oil, omega-3 fatty acids, or any other anti-inflammatory, antithrombotic or anticoagulant agent in the last week
* History of adverse reactions to e-cigarettes

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in measure of platelet aggregometry | 1 Day
  Platelet aggregation is part of the sequence of events leading to the formation of a thrombus (clot).
Change in Measure of Flow Cytometry | 1 Day
  P-Selectin PAC-1 Platelet-Monocyte Aggregates
Change in measure of Endothelial Function Assessment | 1 Day
  Brachial artery flow mediated dilatation (BA-FMD)
Change in measure of Inflammatory Marker Luminex panel-HS-CRP | 1 Day
Change in measure of Inflammatory Marker Luminex panel- IL-6 | 1 Day
Change in measure of Inflammatory Marker Luminex panel- IL-8 | 1 Day
Change in measure of Inflammatory Marker Luminex panel- IL-10 | 1 Day
Change in measure of Inflammatory Marker IL-1b | 1 Day
Change in measure of Inflammatory Marker- endothelin | 1 Day
Change in measure of Inflammatory Marker- TNF-a | 1 Day
Change in measure of Inflammatory Marker- vWF | 1 Day
Change in measure of Inflammatory Marker- thrombomodulin | 1 Day
Change in measure of Inflammatory Marker- E-selectin | 1 Day
Change in measure of Inflammatory Marker- PAI-1 | 1 Day
Change in brachial artery flow mediated dilatation measured non-invasively with a ultrasound probe at rest and after inflation of a forearm blood pressure cuff to 50 mm Hg above measured systolic blood pressure for 5 minutes | 1 Day
Change in blood pressure measured with an automated blood pressure instrument | 1 Day
Change in heart rate measured with an automated blood pressure instrument | 1 Day
Change in pulse oxymetry measured with a pulse oximeter attached to the finger | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — New York University Medical School; Leon H Alviar, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States